CLINICAL TRIAL: NCT04719923
Title: Gut Microbiota, Nutrition and Adverse Reactions to Food in Children With Autism Spectrum Disorders
Brief Title: Dietetic Pattern in Children With Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Associate Professor - Chief of the Pediatric Allergy Program at the Department of Translational Medical Science Chief of the ImmunoNutritionLab at CEINGE - Advanced Biotechnologies, Federico II University
Other Study IDs: 312/17
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with autism spectrum disorders: Children affected by autism spectrum disorders
  Interventions: Behavioral: Children with autism spectrum disorders
- Healthy controls: Healthy children

INTERVENTIONS:
Behavioral: Children with autism spectrum disorders — Subjects affected by autism spectrum disorders
  Groups: Subjects with autism spectrum disorders

SUMMARY:
To date, it is well documented that the gut microbiota (GM) influences numerous physiological processes in the healthy "host". The alteration of the composition and function of the intestinal microbiota, commonly referred to as "dysbiosis", is associated with many pathological conditions. The high co-morbidity between inflammatory bowel diseases and psychiatric symptoms such as anxiety and stress and the frequent presence of gastrointestinal dysfunctions in autistic patients have highlighted a possible implication of GM in psychiatric disorders. The ability of GM to communicate with the central nervous system and the possible influence on behavior led to the discovery of the existence of a microbiota-gut-brain axis. Clinical and experimental data suggest a possible role of modifications in the composition and function of the intestinal microbiota (impaired production of short-chain fatty acids, SCFAs) in major psychiatric disorders such as autism spectrum disorders (ASD). ASD is a severe neurological condition characterized by severe stereotypical behaviors and deficits in linguistic and social interaction. The prevalence of ASD in children is continuously increasing in Western countries. The pathogenesis of ASD is still poorly defined. The clinical manifestations of ASD are the result of complex interactions between genetic, epigenetic, environmental and microbiological factors. The improvement in gastrointestinal symptoms of autistic patients after short-term oral treatment with antibiotics and probiotics clearly indicated a role of the metabolites of MI in ASD. In particular, an alteration in the phyla of Bacteroidetes and Firmicutes in fecal samples from autistic children has been described with conflicting results. Williams and colleagues (2011) evaluated a significant increase in the Firmicutes / Bacteroidetes ratio in intestinal biopsies of autistic children with gastrointestinal disorders. It has also been shown in animal models of ASD that dysbiosis is positively associated with an increase in butyrate levels and inversely associated with the "score" of the severity of ASD symptoms. Alterations in nutritional status, eating habits and adverse reactions to food appear to be more frequent in children with ASD. Several studies support the hypothesis that children with ASD have a greater refusal of food, requiring specific food presentations or eating a reduced variety of foods compared to children without ASD. These conditions are associated with dysbiosis. Preliminary data suggest that particular elimination diets and / or modifications of the intestinal microbiota can determine a positive effect on the symptoms of ASD. A better knowledge of the composition and functions of the intestinal microbiota also in relation to eating habits and the presence of adverse reactions to food in the child with ASD could facilitate new effective strategies for the prevention and treatment of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* subjects with diagnosis Autism Spectrum Disorder or healthy controls

Exclusion Criteria:

* Concomitant presence of:
* epilepsy
* neurological syndromes,
* immunodeficiencies,
* type 1 diabetes
* endocrine diseases,
* congenital heart disease,
* inborn errors of metabolism,
* tuberculosis,
* cystic fibrosis,
* chronic tract diseases respiratory,
* malignancy,

  •Major malformations
* previous surgeries of the gastrointestinal / urinary / respiratory tract
* Use of antibiotics or anti-mycotic and / or pre / pro / synbiotics during the 12 weeks prior to enrollment.
* investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.

Ages: 18 Months to 7 Years | Sex: All
Age Groups: Child
Study Population: 200 subjects of both sexes diagnosed with Autism Spectrum Disorder (ASD),aged between 18 months and 7 years, consecutively observed in the care facility of the Department of Translational Medical Sciences, University of Naples "Federico II" or healthy controls (100/group)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Adverse food reactions | at enrollment
  The evaluation of the occurrence of food reaction is study population

SECONDARY OUTCOMES:
Eating habits | at the entrollment
  The evaluation of eating habits with the 3-day food diary
Nutritional status | at the entrollment
  The evaluation of nutritional status with the collection of auxological data
Composition of gut microbiota | at the entrollment
  The evaluation of intestinal microbiota with the shotgun analysis
Function of gut microbiota | at enrollment
  The evaluation of short chain fatty acids with the gascromatography

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

REFERENCES:
- [Derived] Coppola S, Nocerino R, Oglio F, Golia P, Falco MC, Riccio MP, Carucci L, Rea T, Simeone S, Garotti R, Marani N, Bravaccio C, Canani RB. Adverse food reactions and alterations in nutritional status in children with autism spectrum disorders: results of the NAFRA project. Ital J Pediatr. 2024 Nov 4;50(1):228. doi: 10.1186/s13052-024-01794-8. PMID 39497088